CLINICAL TRIAL: NCT03372941
Title: Hospital Avoidance Strategies for Treatment of Acute Bacterial Skin and Skin Structure Infection (ABSSSI)
Brief Title: Hospital Avoidance Strategies for ABSSSI
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding and recruitment limited by pandemic
Sponsor: Washington University School of Medicine (Other)
Collaborators: The Foundation for Barnes-Jewish Hospital (Other); Allergan (Industry)
Responsible Party: Principal Investigator, Stephen Liang, Principal investigator, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201709136
Record Dates: First submitted 2017-12-04; First posted 2017-12-14 (Actual); Results first posted 2022-12-09 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-11

CONDITIONS: Skin Infection
Keywords: Acute bacterial skin and skin structure infections; Hospital avoidance; Antibiotic therapy; Dalbavancin; Emergency department
MeSH Terms: conditions — Cellulitis; Emergencies | interventions — dalbavancin

STUDY DESIGN:
Intervention Model Description: This study will be single center, randomized, non-blinded study comparing two active treatment arms to treat uncomplicated ABSSSI suspected to be due to Gram-positive bacteria:
  * Alternative treatment strategy comprised of a single dose of dalbavancin administered in the BJH ED or ED observation unit followed by discharge w/ close Infectious Disease outpatient clinic follow-up vs.
  * "Usual care" (i.e., hospital admission for intravenous antibiotics - typically, vancomycin) - antibiotic and doses to be determined at the discretion of the treating clinician (both in the BJH ED and on the BJH inpatient ward)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Alternative treatment strategy (Active Comparator): Patient will receive a single dose of dalbavancin administered in the BJH ED or ED observation unit for ABSSSI followed by discharge w/ close Infectious Disease outpatient clinic follow-up.
  Interventions: Drug: Dalbavancin
- Usual care (No Intervention): Patients will receive "usual care" (i.e., hospital admission for intravenous antibiotics - typically, vancomycin) - antibiotic and doses to be determined at the discretion of the treating clinician (both in the BJH ED and on the BJH inpatient ward).

INTERVENTIONS:
Drug: Dalbavancin — Dalbavancin, a lipoglycopeptide antibiotic, has been approved by the FDA for the treatment of ABSSSI caused by Gram-positive bacteria. A single dose of dalbavancin will be administered in the Emergency Department followed by discharge with close outpatient infectious disease clinic follow-up.
  Other Names: Dalvance
  Arms: Alternative treatment strategy

SUMMARY:
More than 40% of patients presenting with acute bacterial skin and skin structure infection (ABSSSI) to the Barnes-Jewish Hospital (BJH) emergency department (ED) are admitted for intravenous antibiotics. There is growing evidence to suggest that many hospital admissions for uncomplicated ABSSSI due to Gram-positive bacteria could be avoided with an alternative treatment strategy employing newer long-acting antibiotics. Coupled with close outpatient follow-up, such an alternative hospital avoidance strategy has the potential to improve quality and value of care for patients with uncomplicated ABSSSI and optimize use of limited inpatient healthcare resources.

DETAILED DESCRIPTION:
This study seeks to establish the feasibility and acceptability of an alternative treatment strategy for uncomplicated acute bacterial skin and skin structure infection (ABSSSI) in the Barnes Jewish Hospital (BJH) Emergency Department (ED) focusing on hospital admission avoidance using single-dose, long-acting antimicrobial therapy complemented by close follow-up in the ambulatory setting. The extended half-life of these new antimicrobials (dalbavancin, oritavancin) allows for an effective treatment course of >7 days with a single dose, which is the accepted duration for which ABSSSI is usually treated with daily doses of other intravenous or oral antimicrobials. The investigators believe that such an approach will conserve hospital resources by reducing admissions for uncomplicated ABSSSI while delivering comparable if not superior care for this disease, allowing optimal utilization of BJH inpatient beds for other serious medical conditions requiring inpatient care. The investigators believe this novel alternative approach will allow hospitals such as BJH to more cost-effectively and efficiently manage ABSSSI patients. This study will reduce the number of >2 midnight observation admissions to BJH for ABSSSI, thereby improving inpatient capacity to care for patients requiring >2 midnight hospital inpatient admission.

The investigators will conduct a randomized controlled trial comparing patients treated with a single-dose of intravenous dalbavancin (an antibiotic that has been FDA-approved for the treatment of ABSSSI and is currently being used in clinical practice in the U.S.) and discharged home from the ED with close ambulatory care follow-up in clinic vs. patients treated with "usual care" (hospital admission for multiple doses of intravenous vancomycin or other antibiotic directed towards Gram-positive bacteria). Clinical outcomes, healthcare utilization, hospital costs, and patient satisfaction will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age ≥18 years)
* Diagnosis of uncomplicated ABSSSI suspected to be due to Gram-positive bacteria by treating ED clinician, with presence of the following:

  1. Skin lesion size ≥75 cm2 (measured by area of erythema, edema, and/or induration) AND
  2. Signs of systemic inflammation (at least 1 of the following: WBC >12,000 or <4,000 cells/mm3; ≥10% immature neutrophils on peripheral smear; temperature >38.3˚C or <36˚C; heart rate >90 bpm, respiratory rate >20 bpm). Signs of systemic inflammation not required if the patient is age >70 years, has diabetes mellitus, or has been treated with immunosuppressive or chemotherapy in the past 90 days.
* Clinical determination by treating ED clinician that patient will need hospital admission for the sole purpose of receiving intravenous antibiotics directed only towards Gram-positive bacteria (e.g., vancomycin, cefazolin) to treat uncomplicated ABSSSI

Exclusion Criteria:

* Risk for ABSSSI due to Gram-negative bacteria (neutropenia with absolute neutrophil count <500 cells/µL, HIV or severely immunocompromised, burns, infection after trauma or as a result of an aquatic environment, infection after skin graft)
* Any abscess requiring bedside or operative drainage
* Infection due to a vascular catheter or prosthetic device
* Infection of a diabetic foot ulcer or decubitus ulcer
* Necrotizing soft tissue infection
* Sepsis (quick SOFA score ≥2) or septic shock (requiring vasopressors to maintain mean arterial pressure ≥65 mmHg despite resuscitation with at least 30mL/kg of IV crystalloid within first 3 hours)
* Recent antibiotics in prior 14 days
* Hypersensitivity to glycopeptides (vancomycin, televancin, dalbavancin, oritavancin)
* Severe renal insufficiency (CrCl <30 mL/min)
* Severe hepatic insufficiency (Child-Pugh Class C)
* Pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2021-10-14 (Actual); Study Completion 2021-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Y Liang, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Barnes-Jewish Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Alternative Treatment Strategy | Usual Care
Started | 6 | 5
Completed | 4 | 1
Not Completed | 2 | 4
Not completed — Lost to Follow-up | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alternative Treatment Strategy | Usual Care | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Continuous [Mean (Full Range); unit: years] | 43.3 [29 to 55] | 42.4 [21 to 71] | 42.9 [21 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 4 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 3 | 1 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Healthcare Utilization Related to ABSSSI
Description: Repeat ED visit(s) within 28 days, need for hospital admission(s) to receive intravenous antibiotics ("alternative treatment strategy" arm), or need for switch to different oral or intravenous antibiotic to treat ABSSSI ("usual care" arm)
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Alternative Treatment Strategy | Usual Care
Number analyzed (Participants) | 6 | 5
Participants
  Number of participants with repeat ED visit | 0 | 1
  Number of participants with need for hospital admission(s) to receive IV antibiotics | 1 | 0
  Number of patients without additional healthcare utilization to treat ABSSSI | 5 | 4
  Number of participants with need for switch to different oral antibiotic | 0 | 0

2. Secondary Outcome: Healthcare Cost Related to ABSSSI Management
Description: Indirect/direct costs associated with ED visit(s), indirect/direct costs associated with hospital admission(s)
Time Frame: 28 days
Population: Data were not collected
Arm/Group | Alternative Treatment Strategy | Usual Care
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Clinical Response
Description: Change in ABSSSI lesion area (cm2)
Time Frame: 28 days
Population: Data were not collected
Arm/Group | Alternative Treatment Strategy | Usual Care
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Clinical Success
Description: Clinical resolution of symptoms, need for additional intravenous/oral antibiotic therapy
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Alternative Treatment Strategy | Usual Care
Number analyzed (Participants) | 4 | 1
Participants
  Number of participants with clinical resolution of symptoms | 4 | 1
  Number of participants with need for additional intravenous/oral antibiotic therapy | 0 | 0

5. Secondary Outcome: Overall Patient Satisfaction Based on Standardized Measures
Description: Hospital Consumer Assessment of Healthcare Providers and Systems (HCAHPS) survey items
Time Frame: 28 days
Population: Data were not collected
Arm/Group | Alternative Treatment Strategy | Usual Care
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Patient Satisfaction Specific to ABSSSI Care
Description: Targeted survey questions specific to ABSSSI and patient-centered outcomes with relation to alternative treatment strategy vs. usual care
Time Frame: 28 days
Population: Data were not collected
Arm/Group | Alternative Treatment Strategy | Usual Care
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Patient Safety
Description: Adverse drug events
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Alternative Treatment Strategy | Usual Care
Number analyzed (Participants) | 4 | 1
Participants
  Number of participants with an adverse drug event | 0 | 0
  Number of participants without an adverse drug event | 4 | 1

8. Secondary Outcome: Quality of Life Measured Using RAND SF-36 Survey
Description: RAND SF-36
Time Frame: 28 days
Population: Data were not collected
Arm/Group | Alternative Treatment Strategy | Usual Care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Alternative Treatment Strategy | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 0/6 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-28): https://cdn.clinicaltrials.gov/large-docs/41/NCT03372941/Prot_SAP_000.pdf